CLINICAL TRIAL: NCT06573957
Title: Comparison of the Effects of Intravenous Administration of Dexmedetomidine 0.5 μg/kg Body Weight With Intravenous Lidocaine 1.5 mg/kg Body Weight on Blood Pressure and Heart Rate Response During Laryngoscopy and Endotracheal Intubation
Brief Title: Comparison of the Effects of Dexmedetomidine and Lidocaine on Blood Pressure and Heart Rate Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AN-202408.01
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: General Anesthesia
Keywords: Haemodynamic Response; Endotracheal Intubation; Dexmedetomidine; Lidocaine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Twenty-one patients are administered dexmedetomidine at a dose of 0.5 µg/kg body weight 10 minutes before induction, then receive general anesthesia induction with intravenous propofol 2 mg/kg body weight and intravenous atracurium 0.5 mg/kg body weight. Positive pressure ventilation is then applied for 3 minutes using a ventilator in volume control mode with a tidal volume of 6-8 mL/kg body weight, a respiratory rate of 12 breaths per minute, and PEEP 5. Oxygen at 3 liters, air at 3 liters, and sevoflurane at 2 vol% are set.
  Interventions: Drug: Dexmedetomidine
- Lidocaine (Active Comparator): Twenty-one patients receive general anesthesia induction with intravenous propofol 2 mg/kg body weight and intravenous atracurium 0.5 mg/kg body weight. Positive pressure ventilation is then applied for 3 minutes using a ventilator in volume control mode with a tidal volume of 6-8 mL/kg body weight, a respiratory rate of 12 breaths per minute, and PEEP 5. Oxygen at 3 liters, air at 3 liters, and sevoflurane at 2 vol% are set, followed by lidocaine at 1.5 mg/kg body weight in a 5cc syringe 90 seconds before intubation.
  Interventions: Drug: Lidocain

INTERVENTIONS:
Drug: Dexmedetomidine — Patient in experimental arms will received intravenous dexmedetomidine at a dose of 0.5 µg/kg body weight 10 minutes before general anesthesia induction
  Arms: Dexmedetomidine
Drug: Lidocain — Patient in experimental arms will receive intravenous lidocaine at 1.5 mg/kg body weight in a 5cc syringe 90 seconds before intubation
  Arms: Lidocaine

SUMMARY:
Endotracheal intubation is considered a definitive therapy and the gold standard for airway management. However, this procedure carries several risks, including sudden increases in blood pressure and heart rate. These spikes in blood pressure and heart rate can be tolerated by healthy individuals, but for patients with cerebrovascular and cardiovascular risk factors, they can be extremely dangerous and even life-threatening. Various techniques and drug choices can be employed to prevent the hemodynamic surges associated with endotracheal intubation, including the use of anesthetic drugs from the α2-adrenergic agonist and amide classes. One of the α2-adrenergic agonists commonly used to prevent hemodynamic surges during endotracheal intubation is dexmedetomidine, while one of the amide drugs frequently used for this purpose is lidocaine.

DETAILED DESCRIPTION:
Dexmedetomidine works very selectively on noradrenergic receptors distributed both within and outside the central nervous system, particularly in the pons and medulla. Presynaptic stimulation of α2 receptors can reduce the release of norepinephrine and the activation of postsynaptic α2 receptors. Lidocaine works by inhibiting sodium channels within cells, preventing the occurrence of action potentials and the transmission of impulses along nerves. Lidocaine also acts by blocking calcium and potassium channels as well as N-methyl-D-aspartate (NMDA) receptors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-59 years.
* Patients scheduled for oral intubation.
* Physical status ASA I and II (American Society of Anesthesiologists).
* Patients with Mallampati classification I-II.

Exclusion Criteria:

* History of allergy to the drugs that will be used.
* Pregnant patients.
* Patients taking medications that affect blood pressure and heart rate, such as vasodilators, adrenergic blockers, antiarrhythmics, and cardiac stimulants.
* Patients with arrhythmias, AV block, liver disorders, hypertension, and hypoalbuminemia.
* Patients who have been given opioids within the last 24 hours.
* Patients with predicted intubation difficulties.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Right after endotracheal intubation until 5 minutes after endotracheal intubation
Diastolic blood pressure | Right after endotracheal intubation until 5 minutes after endotracheal intubation
Heart rate | Right after endotracheal intubation until 5 minutes after endotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP Dr. Hasan Sadikin, Bandung, West Java, Indonesia